CLINICAL TRIAL: NCT05476562
Title: Real-World Treatment Patterns, Healthcare Resource Utilization and Associated Costs Among Patients With Chronic Myeloid Leukemia in Later Lines of Therapy
Brief Title: Study Conducted Among Patients With CML
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001AUS07
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukemia,; tyrosine kinase inhibitors,; treatment patterns,; HRU,; costs
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Tyrosine Kinase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- First-line Therapy: A cohort of adult patients with CML who were treated with TKIs were identified using the IBM® MarketScan® Commercial and Medicare Supplemental databases (commercial claims; the MarketScan database)
  Interventions: Other: Tyrosine Kinase Inhibitors (TKIs)
- Second-line Therapy: A cohort of adult patients with CML who were treated with TKIs were identified using the IBM® MarketScan® Commercial and Medicare Supplemental databases (commercial claims; the MarketScan database)
  Interventions: Other: Tyrosine Kinase Inhibitors (TKIs)
- Third-line Therapy: A cohort of adult patients with CML who were treated with TKIs were identified using the IBM® MarketScan® Commercial and Medicare Supplemental databases (commercial claims; the MarketScan database)
  Interventions: Other: Tyrosine Kinase Inhibitors (TKIs)
- Fourth-line Therapy: A cohort of adult patients with CML who were treated with TKIs were identified using the IBM® MarketScan® Commercial and Medicare Supplemental databases (commercial claims; the MarketScan database)
  Interventions: Other: Tyrosine Kinase Inhibitors (TKIs)

INTERVENTIONS:
Other: Tyrosine Kinase Inhibitors (TKIs) — The study included patients with CML who were previously treated with TKIs, who are relapsed/refractory to/intolerant of TKIs on third or later lines of therapy in the US.

SUMMARY:
Retrospective, non-interventional observational cohort study conducted among patients with CML.

DETAILED DESCRIPTION:
A retrospective, non-interventional cohort study was used to address the study objectives. A cohort of adult patients with CML who were treated with TKIs were identified using the IBM® MarketScan® Commercial and Medicare Supplemental databases (commercial claims; the MarketScan database) to have a better understanding of real-world treatment patterns, HRU and healthcare costs among patients with CML treated with later lines of therapy (i.e., third line or later).

For Phase I, the IBM® MarketScan® Commercial Claims and Encounters and Medicare Supplemental Databases were used (commercial claims). The commercial claims covered the period from 01/01/2001 to 06/30/2019.

The study consisted of the following periods:

* The baseline period was defined as the 6-month period before the first line therapy initiation for CML.
* The observation period was defined as the period of at least 12 months from the first CML diagnosis to the end of data availability or end of health plan coverage, whichever occurs first; the observation period varied by patient.

ELIGIBILITY:
Inclusion Criteria:

Patients were selected for the analysis of later lines of therapy in commercial claims (i.e., were previously treated with TKIs, who are relapsed/refractory to/intolerant of TKIs) if they met the following criteria:

* Had at least one diagnosis for CML, with first CML diagnosis observed in claims on or after May 10, 2001, the date of FDA approval for imatinib
* Were at least 18 years of age as of the first CML diagnosis
* Started a first line therapy for CML with imatinib, dasatinib, nilotinib, or bosutinib (conditional on FDA-approval dates)
* Initiated first line therapy within a maximum of 1 month prior to the first diagnosis for CML or a maximum 3 months following the first diagnosis for CML
* Had continuous health plan enrollment (pharmacy and medical benefits) from the washout period to at least 12 months following the first CML diagnosis

Exclusion Criteria:

* Patients had a diagnosis for CML remission or relapse anytime prior to first line therapy
* Patients had a medical claim associated with a clinical trial during the washout period up to the end of the observation period
* Patients had an HSCT during the washout period up to the first line therapy initiation
* Patients had chemotherapy treatment (except hydroxyurea) during the washout period up to the first line therapy initiation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted among patients with CML.
Sampling Method: Non-Probability Sample
Enrollment: 3234 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Number of patients across all lines of therapy | throughout the study, approximately 20 years
  Number of patients across all lines of therapy were reported to evaluate treatment sequences among the patients.
Number of patients with the use of pre-treatment hydroxyurea | throughout the study, approximately 20 years
  Number of patients with the use of pre-treatment hydroxyurea were reported to evaluate treatment patterns in patients.
Number of patients Treatment received and initial dose at each line | throughout the study, approximately 20 years
  Number of patients Treatment received and initial dose at each line were reported to evaluate treatment patterns in patients.
Number of patients as per the calendar year of line of therapy initiation | throughout the study, approximately 20 years
  Number of patients as per the calendar year of line of therapy initiation were reported to evaluate treatment patterns in patients.
Duration of the line of therapy | throughout the study, approximately 20 years
  Duration of the line of therapy was reported to evaluate treatment patterns in patients.
Treatment-free period among those with an observed subsequent line of therapy | throughout the study, approximately 20 years
  Treatment-free period among those with an observed subsequent line of therapy was reported to evaluate treatment patterns in patients.
Number of patients who discontinued treatment | throughout the study, approximately 20 years
  Number of patients who discontinued treatment were reported to evaluate treatment patterns in patients.
Number of patients: All cause Health Resource Utilization among patients with three lines of therapy or more | throughout the study, approximately 20 years
  Number of patients: All cause Health Resource Utilization were reported to estimate HRU among patients with three lines of therapy or more.
Healthcare costs among patients with three lines of therapy or more | throughout the study, approximately 20 years
  Healthcare costs among patients with three lines of therapy or more were reported.

SECONDARY OUTCOMES:
Prevalence of second and third or later lines of therapy | Calendar year 2006 to 2018, approximately 12 years
  Prevalence was defined as the number of cases alive per year of patients with CML who were currently or previously treated on later lines of therapy (third line or later), by calendar year from 2006 to 2018
Healthcare costs among patients with earlier lines of therapy | throughout the study, approximately 20 years
  Healthcare costs among patients with earlier lines of therapy were reported.
Number of patients: All cause Health Resource Utilization among patients with earlier lines of therapy | throughout the study, approximately 20 years
  Number of patients: All cause Health Resource Utilization among patients with earlier lines of therapy were reported.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CABL001AUS07 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17964